CLINICAL TRIAL: NCT02211833
Title: A Phase I Open-label Dose Escalation Study of Intravenous BI 2536 Together With Pemetrexed in Previously Treated Patients With Non-small-cell Lung Cancer
Brief Title: Dose Escalation Study of BI 2536 With Pemetrexed in Previously Treated Patients With Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1216.5
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BI 2536; Pemetrexed

ARMS (1):
- BI 2536 with pemetrexed (Experimental): combination therapy phase may be followed by BI 2536 monotherapy for eligible patients
  Interventions: Drug: BI 2536; Drug: Pemetrexed

INTERVENTIONS:
Drug: BI 2536
Drug: Pemetrexed

SUMMARY:
Exploratory evaluation of safety, tolerability, pharmacokinetics (PK), maximum tolerated dose (MTD), and efficacy of BI 2536 administered in combination with pemetrexed

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic or cytologic confirmed diagnosis of NSCLC
2. Recurrent, advanced or metastatic NSCLC that had progressed following 1 prior chemotherapy regimen for advanced disease. Patients could have received prior adjuvant chemotherapy as long as the disease free interval was longer than 1 year.
3. Measurable disease by 1 or more techniques (CT, MRI) according to RECIST criteria
4. Male or female aged 18 years or older
5. Life expectancy of at least 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance score 0-2
7. Written informed consent that was consistent with International Conference on Harmonization (ICH) - Good Clinical Practice (GCP) guidelines

Exclusion Criteria:

1. Treatment with an investigational drug in another clinical study within the 28 days prior to the start of therapy or concomitantly with this study
2. Anti-cancer therapy for NSCLC (except radiotherapy for palliative reasons) within the 28 days prior to Day 1 of treatment period 1 of this trial
3. Any persisting toxicities that were deemed to be clinically significant from the previous therapy
4. Received more than 1 prior chemotherapy regimen for advanced disease (not including prior adjuvant therapy). Patients could have received prior epidermal growth factor receptor tyrosine kinase inhibitors
5. Unwilling or unable to take folic acid and vitamin B12 supplementation
6. Active brain metastases (stable for <28 days, symptomatic, or requiring concurrent steroids). Patients who had received prior whole brain irradiation and whose brain metastases were stable according to the criteria above were not excluded
7. Other active malignancy diagnosed within the past 3 years (other than non-melanomatous skin cancer and cervical intraepithelial neoplasia)
8. Concomitant intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would have limited compliance with trial requirement or which were considered relevant for the evaluation of the efficacy or safety of the trial drug
9. Unable or unwilling to interrupt concomitant administration of NSAIDS 5 days prior to the day of and up to 2 days after the administration of pemetrexed
10. Received prior therapy with pemetrexed
11. Absolute neutrophil count (ANC) ≤1 500/μL, platelet count ≤100 000/μL, or haemoglobin <9 mg/dL
12. Total bilirubin >1.5 mg/dL (26 μmol/L), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥2.5 x the upper limit of normal (ULN), except in cases of known liver metastasis where a maximum 5 x ULN was acceptable
13. Serum creatinine level >1.5 mg/dL and or creatinine clearance <45 mL/min
14. Sexually active and unwilling to use a medically acceptable method of contraception
15. Pregnancy or breast feeding
16. Known or suspected active alcohol or drug abuse
17. Unable to comply with the protocol
18. Any known hypersensitivity to the trial drugs or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BI 2536 in combination with pemetrexed | up to 3 weeks
  by occurrence of dose limiting toxicities (DLT)
Number of patients with adverse events during combination therapy | up to 20 weeks
  according to common terminology criteria for adverse events (CTCAE) 3.0

SECONDARY OUTCOMES:
Objective tumor response after combination therapy | up to 20 weeks
  according to Response Evaluation Criteria in Solid Tumours (RECIST)
Duration of objective tumor response after combination therapy | up to 1 year
Progression free survival (PFS) | up to 2 years
Overall survival | up to 2 years
Number of patients with abnormal laboratory findings | up to 20 weeks
Change in Eastern Cooperative Oncology Group (ECOG) performance score | baseline, up to 1 year